CLINICAL TRIAL: NCT02175576
Title: Randomized Controlled Clinical Outcomes of the Vanguard XP Bicruciate Knee System
Acronym: GK9B
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data no longer required to meet regulatory requirements.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTHO.CR.GK9B
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Lower Limb Deformity; Post-traumatic Deformity; Complications, Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vanguard XP Bicruciate Knee System (Experimental): 153 patients receive Vanguard XP Bicruciate Knee System
  Interventions: Device: Vanguard XP Bicruciate Knee System
- Vanguard CR Knee System (Active Comparator): 153 patients receive Vanguard CR Knee System
  Interventions: Device: Vanguard CR Knee System

INTERVENTIONS:
Device: Vanguard XP Bicruciate Knee System — The Vanguard XP is a bicruciate retaining total knee design and is constrained by natural soft tissue.
  Arms: Vanguard XP Bicruciate Knee System
Device: Vanguard CR Knee System — The Vanguard CR system requires the ACL to be sacrificed and is constrained by soft tissue and device design.
  Arms: Vanguard CR Knee System

SUMMARY:
Randomized Controlled Study to determine if preservation of ligaments provides increased functional ability post-operatively in comparison to traditional TKA which sacrifices soft tissue.

DETAILED DESCRIPTION:
Randomized Controlled Study to compare clinical and patient reported outcomes of the Vanguard XP Bicruciate Total Knee System to the Vanguard CR Knee System through 10 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* cemented application of components
* bilateral subjects randomized by knee
* patients with pre-existing contralateral knee surgery
* painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, or traumatic arthritis where one or more compartments are involved
* correction of varus, valgus, or posttraumatic deformity
* sufficient soft tissue surrounding the knee, including the Anterior Cruciate Ligament

Exclusion Criteria:

* cementless application of components
* BMI greater than or equal to 40
* use of Anterior Stabilized Bearings
* patients with severe pre-operative varus or valgus deformity greater than or equal to 15 degrees
* correction or revision of previous joint replacement procedure on index knee
* infection
* sepsis
* osteomyelitis

Relative exclusion criteria:

* uncooperative patient or patient with neurological disorders who is incapable of following directions
* osteoporosis
* metabolic disorders which may impair bone formation
* osteomalacia
* distant foci of infections which may spread to the implant site
* rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* vascular insufficiency, muscular atrophy, neuromuscular disease
* incomplete or deficient soft tissue surrounding the knee, including the anterior cruciate ligament

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (2):
- United States (2):
  - Midwest Orthopaedics at Rush University Medical Center, Chicago, Illinois
  - University of Utah Orthopaedic Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After obtaining informed consent, participants were evaluated according to protocol-defined eligibility (inclusion and exclusion) criteria. If a participant did not meet the eligibility criteria, he or she was excluded from participation and not assigned to a study group.
Units Other Than Participants: Knees
Period: Overall Study
Arm/Group | Vanguard XP Bicruciate Knee System | Vanguard CR Knee System
Started | 20; 22 Knees (Two (2) participants enrolled both knees into the study.) | 30; 33 Knees (Three (3) participants enrolled both knees into the study.)
12 Month Follow-Up Visit (Participants for which the primary endpoint of Modified Knee Society Score (mKSS) at 12 months could be analyzed.) | 8; 10 Knees | 18; 21 Knees
Completed | 0; 0 Knees (Study was terminated prior to reaching the final follow-up visit as described in the protocol.) | 0; 0 Knees (Study was terminated prior to reaching the final follow-up visit as described in the protocol.)
Not Completed | 20; 22 Knees | 30; 33 Knees

BASELINE CHARACTERISTICS:
Units Other Than Participants: Knees
Groups:
- Total: Total of all reporting groups
Arm/Group | Vanguard XP Bicruciate Knee System | Vanguard CR Knee System | Total
Number analyzed (Participants) | 20 | 30 | 50
Number analyzed (Knees) | 22 | 33 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.0) | 66.4 (7.3) | 65.5 (7.6)
Sex: Female, Male [Count of Units; unit: Knees]
  Female | 13 | 17 | 30
  Male | 9 | 16 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 30 | 50
Modified Knee Society Score [Mean (Standard Deviation); unit: score on a scale] — The American Knee Society Score is part clinical exam and part patient administered assessment of the knee. The objective part of the score was collected in the clinic by qualified personnel. The functional and pain components of the score were collected by patient completed questionnaire. Total scores can range from 0 to 200, with higher scores indicating better outcomes.
  score on a scale | 111.0 (27.0) | 114.5 (27.6) | 113.1 (27.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Knees Reported as "Feels Normal" on a Single Assessment Numeric Evaluation (SANE)
Description: Participants answered a Single Assessment Numeric Evaluation (SANE) which asked how they rated their knee function. A score of 100 indicates normal and anything below 100 indicates a percentage of normal function.
Time Frame: 12 Months
Population: All knees that contributed a SANE score for function at 12 months were included in the analysis.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Vanguard XP Bicruciate Knee System | Vanguard CR Knee System
Number analyzed (Participants) | 12 | 20
Number analyzed (Knees) | 14 | 23
Knees | 1 | 2

2. Secondary Outcome: Modified Knee Society Score
Description: The American Knee Society Score is part clinical exam and part patient administered assessment of the knee. The objective part of the score was collected in the clinic by qualified personnel. The functional and pain components of the score were collected by patient completed questionnaire. Total scores can range from 0 to 200, with higher scores indicating better outcomes.
Time Frame: 12 months
Population: All patients that contributed a Modified Knee Society Score (mKSS) at 12 months were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Knees
Arm/Group | Vanguard XP Bicruciate Knee System | Vanguard CR Knee System
Number analyzed (Participants) | 8 | 18
Number analyzed (Knees) | 10 | 21
score on a scale | 164.6 (29.4) | 168.7 (30.9)

3. Secondary Outcome: Revisions/Removals
Description: Number of study device revisions or removals reported during the study.
Time Frame: 3 years
Population: Participants who were randomized, underwent surgery, and received the study device.
Measure: Number; unit: Revisions/Reoperations
Arm/Group | Vanguard XP Bicruciate Knee System | Vanguard CR Knee System
Number analyzed (Participants) | 20 | 30
Revisions/Reoperations | 0 | 0

4. Secondary Outcome: Number of Knees Reported as "Feels at Least 80% of Normal" on a Single Assessment Numeric Evaluation (SANE)
Description: as for outcome 1
Time Frame: 12 Months
Population: All knees that contributed a SANE score for function at 12 months were included in the analysis.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Vanguard XP Bicruciate Knee System | Vanguard CR Knee System
Number analyzed (Participants) | 12 | 20
Number analyzed (Knees) | 14 | 23
Knees | 10 | 20

5. Secondary Outcome: Number of Knees With Which Participants Reported Being "Happy" or "Very Happy"
Description: Participants answered a survey which asked how they they would describe their satisfaction with their new joint. Options for answers included "I have never been happy," "Ok - but not perfect," "Happy," and "Very Happy."
Time Frame: 12 Months
Population: All patients that contributed a patient satisfaction score at 12 months were included in the analysis.
Measure: Count of Units; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Vanguard XP Bicruciate Knee System | Vanguard CR Knee System
Number analyzed (Participants) | 12 | 20
Number analyzed (Knees) | 14 | 23
Knees | 12 | 18

ADVERSE EVENTS:
Time Frame: 3 years
Description: Per the study protocol, only device-related and serious adverse events were collected in this study.
Arm/Group | Vanguard XP Bicruciate Knee System | Vanguard CR Knee System
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/30
Serious Adverse Events (participants affected / at risk) | 5/20 | 7/30
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vanguard XP Bicruciate Knee System (N=20) | Vanguard CR Knee System (N=30)
Fracture of patella (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Instability Medial/Lateral (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stiff knee resulting in manipulation (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Effusion/swelling and pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Synvectomy and lysis of adhesions (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sciatic nerve pain (Nervous system disorders) | 1 (1) | 0 (0)
Pain, stiffness, decrease in satisfaction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vanguard XP Bicruciate Knee System (N=1) | Vanguard CR Knee System (N=3)
Radiograph radiolucency seen under tibial platform (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nerve Deficit (Nervous system disorders) | 0 (0) | 1 (1)
Periosteal reaction medial cortex (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Effusion and pain to knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02175576/Prot_SAP_000.pdf